CLINICAL TRIAL: NCT06238531
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase Ib Study to Evaluate the Safety, Tolerability, And Pharmacokinetics of Gusacitinib in Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: A Clinical Trial to Evaluate Safety of Gusacitinib in Patients With Systemic Lupus Erythematosus (SLE) or Lupus
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug company discontinuing study.
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10001700; 001700-AR
Record Dates: First submitted 2024-02-01; First posted 2024-02-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Lupus; Systemic Lupus Erythematosus; Gusacitinib; Investigational Drug; Treatment; Mild
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lymphoma, Follicular | interventions — gusacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Subjects will remain on their usual SLE medications
- Placebo (Placebo Comparator): Subjects will receive a placebo that looks similar to the interventional drug.
  Interventions: Drug: Gusacitinib

INTERVENTIONS:
Drug: Gusacitinib — An orally active dual SYK/JAK kinase inhibitor
  Arms: Placebo

SUMMARY:
Background:

Systemic lupus erythematosus (SLE), also called lupus, is a disease that causes the body s immune system to attack healthy tissue. Lupus causes swelling and inflammation in the skin, skin, joints, kidneys, brain, blood vessels, and other organs. There is no cure for lupus. Current treatments do not help everyone and may have adverse effects. Better treatments are needed.

Objective:

To test a study drug (Gusacitinib) in people with lupus.

Eligibility:

People aged 18 years and older with lupus.

Design:

Participants will be screened. They will have a physical exam with blood and urine tests and a test of their heart function. They will have a chest X-ray. They will have tests that use blood pressure cuffs to measure blood flow and pressure throughout the body.

Participants will have 9 clinic visits and 6 phone visits over about 7 months.

The study has 3 parts.

Part 1: Gusacitinib is a tablet taken by mouth. Participants will be divided into 3 groups. One group will receive the study drug, and a second group will get a placebo. The placebo looks like the study drug but does not contain any medicine. Both of these groups will take their tablets once a day for 12 weeks. The third group will continue to take their usual medications for lupus throughout the study.

Part 2: All participants who took the study drug or placebo in part 1 will take the study drug once a day for 12 weeks.

Part 3: All participants who took the study drug will stop taking it for 4 weeks.

DETAILED DESCRIPTION:
STUDY DESCRIPTION:

This is a phase Ib study of Gusacitinib a dual inhibitor of JAK and SYK kinases, that can simultaneously target multiple signaling pathways responsible for the SLE disease pathogenesis. This study will compare the safety of Gusacitinib 80 mg with placebo initially in a double-blind period and then 80 mg daily in an open label period, followed by an off-drug period.

In addition, we will have a comparator group of SLE subjects receiving standard of care treatment. We hypothesize that Gusacitinib will be safe and well tolerated in subjects with SLE.

OBJECTIVES:

Primary Objective: The primary Objective of the study is to determine safety and tolerability of Gusacitinib 80 mg in subjects with SLE.

Secondary Objectives: Pharmacokinetics of Gusacitinib in SLE. Effects of Gusacitinib on plasma lipid profile, vascular stiffness, and endothelial dysfunction. Efficacy of Gusacitinib in controlling SLE disease activity. Exploratory objectives to understand the effects of dual JAK and SYK inhibition on Interferon Gene Signature, Serum Cytokines, NET formation, and Immune cells phenotype.

ENDPOINTS:

Primary Endpoint: Adverse Events severity (as defined by AEs equal or greater than grade 3 as per the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE) v5.0) and frequency as compared to placebo at week 12.

Secondary Endpoints: Change in the proportion of patients achieving SLE Responder Index-4 (SRI 4) response at week 24 compared to baseline. Another efficacy analysis will be done by comparing subjects treated with Gusacitinib vs. placebo at week 12. SRI-4 response is defined as:

* Reduction of >=4 points from baseline in SLEDAI-2K score
* No new BILAG A or no more than 1 new BILAG B disease activity scores
* No worsening (defined as an increase of >=0.3 points [10 mm] from baseline) in the Physician s Global Assessment of Disease Activity
* Change in SLEDAI-2K total score at week 24

ELIGIBILITY:
* INCLUSION CRITERIA
* Male or female subject, 18 years of age or older, at the time of consent
* Meets at least 4 of 11 modified American College of Rheumatology (ACR) (1997) Revised Criteria for the Classification of Systemic Lupus Erythematosus
* Has no to mild disease activity defined as a SLEDAI 2K score between 0-6.
* If on glucocorticoids, the dose must be prednisone <=20 mg daily (or equivalent) for 2 weeks at the time of screening. At the investigator s discretion, glucocorticoids may be tapered during the second (open label) period of the study.
* If on hydroxychloroquine, the dose must have been stable for the 12 weeks prior to screening visit. The maximum allowed dose is hydroxychloroquine up to 400 mg/day or 6.5 mg/kg/day if more than 400 mg/day; or equivalent dose of other antimalarial medications
* Stable doses of immunosuppressant for the 12 weeks prior to the screening visit. Immunosuppressant medications include azathioprine up to 2 mg/kg, methotrexate up to 20 mg/week, mycophenolate mofetil up to 3000 mg/day or mycophenolic acid <= 2.16 g/day. The subject will be taken off these immunosuppressant medications 2 weeks prior to administration of study medication and will be kept off these medications for the duration of study. Any subject experiencing worsening of SLE disease activity will be treated by a single dose of intra-muscular corticosteroid. This will be allowed only once during each period of the study. A second flare during each period requiring treatment would lead to withdrawal of the subject. The subjects in comparator group will continue on standard of care treatment.
* Stable medications for diabetes, hypertension and/or statins for 12 weeks prior to the screening visit.
* For female subject of childbearing potential involved in any sexual intercourse that could lead to pregnancy: the subject must agree to use a highly effective contraceptive method from at least 4 weeks before Day 1 until at least 4 weeks after the last study product administration. Highly effective contraceptive methods include hormonal contraceptives (e.g. combined oral contraceptive, patch, vaginal ring, injectable, or implant, or progesterone only pill or injections), intrauterine devices or intrauterine systems, vasectomized partner(s), tubal ligation, or double barrier methods of contraception (e.g. male condom with cervical cap, male condom with diaphragm, or male condom with contraceptive sponge) in conjunction with spermicide.

Note: Subjects must have been on a stable dose of hormonal contraceptives for at least 4 weeks before Day 1.

Note: The above list of contraceptive methods does not apply to subjects who are abstinent for at least 4 weeks before Day 1 and will continue to be abstinent from penile-vaginal intercourse throughout the study. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant.

Note: A female subject of nonchildbearing potential is as follows:

* Female subject who has had surgical sterilization (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy);
* Female subject who has had a cessation of menses for at least 12 months without an alternative medical cause, and a follicle-stimulating hormone (FSH) test confirming nonchildbearing potential (as per the reference range of the testing laboratory).

  * For male subject involved in any sexual intercourse that could lead to pregnancy, subject must agree to use one of the highly effective contraceptive methods listed in Inclusion Criterion #8, from Day 1 until at least 90 days after the last study product administration. If the female partner of a male subject use any of the hormonal contraceptive methods listed above, this contraceptive method must be used by the female partner from at least 4 weeks before Day 1 until at least 90 days after the last study product administration by the male subject.
  * Male subjects must not donate sperm from Day 1 until at least 90 days after the last study product administration.
  * Female subject of childbearing potential has had a negative serum pregnancy test at screening and negative urine pregnancy test on Day 1.
  * Subject is willing to participate and can give informed consent.
  * Subjects must be willing to comply with all study procedures and must be available for the duration of the study.

EXCLUSION CRITERIA

An individual who meets any of the following criteria will be excluded from participation in this study:

* Subject is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
* Subject has a history of cancer or lymphoproliferative disease within 5 years prior to Day 1. Note: Subjects with successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix are not to be excluded.
* Subject has any clinically significant medical condition or physical / laboratory / ECG / vital signs abnormality that would, in the opinion of the investigator, put the subject at undue risk or interfere with interpretation of study results.
* Subject has 12-lead ECG abnormalities considered by the investigator to be clinically

significant or a QTcF >= 450 milliseconds, regardless of clinical significance, at screening. Abnormal ECG may be confirmed with one repeated assessment. For subjects with a QTcF >= 450 msec on initial ECG, the mean of the two QTcF values will determine eligibility.

* Subject has congestive heart failure class III or IV as per the New York Heart Association (NYHA) classification.
* Subject has a history of untreated recurrent venous thromboembolic event (VTE) (>= 2 episodes in the past).
* Subject has experienced any of the following within the last 6 months prior to Day 1: VTE, myocardial infarction, angioplasty, or cardiac stent placement, unstable ischemic heart disease, or stroke.
* Subject had other major surgery within 8 weeks prior to Day 1 or has a major surgery planned during the study.
* Subject has positive results for hepatitis B surface antigens (HBsAg), antibodies to hepatitis B core antigens (anti-HBc), hepatitis C virus (HCV), human immunodeficiency virus (HIV), or BK viremia at the screening visit.
* Subject has a known active tuberculosis (TB) or a positive TB infection test. Subject will be evaluated for latent TB infection with a purified protein derivative (PPD) test or a QuantiFERON-TB Gold test. Subjects who demonstrate evidence of latent TB infection (either PPD >= 5 mm of induration or positive QuantiFERON-TB Gold test, irrespective of Bacillus Calmette-Gu(SqrRoot)(Copyright)rin vaccination status) will only be allowed to participate in the study if there is documented evidence of a completed adequate treatment course for latent TB (with negative chest x-ray findings for active TB).
* Subject has a known history of diverticulitis.
* Subject has received any marketed or investigational biologic agent (such as rituximab, belimumab, anifrolumab etc.) within 12 months or 5 half-lives (whichever is longer) prior to Day 1.
* Subject has received a live attenuated vaccine within 4 weeks prior to Day 1 or plans to receive a live attenuated vaccine during the study and up to 4 weeks or 5 half-lives (of the study product), whichever is longer, after the last study product administration.
* Subject has used systemic (Intravenous) antibiotics within 2 weeks prior to Day 1.
* Treatment with cyclophosphamide within the 6 months prior to screening.
* A history of drug or alcohol abuse within the 6 months prior to screening.
* Blood pressure not adequately controlled on the current medications.
* History of chronic liver disease (moderate and severe hepatic impairment (Child-Pugh B and C) or elevated LFTs:

ALT or AST >= 2x upper limit of normal at screening

serum unconjugated bilirubin > 2mg/dL at screening

* Dialysis or serum creatinine >2 mg/dL.
* Protein to creatinine ratio of more than 1000 mg/mg or 24 hours urine protein of more than 1000 mg.
* Active urinary sediment (WBC casts, RBC casts or mixed cellular casts 1+ or more / mcL).
* Hypercholesterolemia: Values after an 8-12 hour fasting blood specimen: total cholesterol >250 mg/dL or LDL >180 mg/dl or hypertriglyceridemia (triglyceride >300 mg/dL) at screening visit.
* Subjects with active renal or central nervous system involvement due to SLE or a BILAG A in any organ system.
* WBC <2500/ L or ANC <1,000/ L, Hgb <9.0 g/dL or platelets <70,000/ L or absolute lymphocyte count < 500/ L at screening and present on repeat testing up to 4 weeks apart
* Current treatment with potent inhibitors of Cytochrome P450 3A4 (CYP3A4) (e.g., ketoconazole) or receiving one or more concomitant medications that result in both moderate inhibition of CYP3A4 and potent inhibition of CYP2C19 (e.g., fluconazole) that would increase serum availability of Gusacitinib. Past treatment with the above mentioned agent is allowed if it was more than a week prior to the administration of the first dose of study medication.
* Current treatment with strong and moderate inhibitors of CYPs 3A4, 2C8, 2D6, and inhibitors of BCRP and MDR1. Past treatment with the above mentioned agent is allowed if it was more than a week prior to the administration of the first dose of study medication.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Adverse Events severity (as defined by AEs equal or greater than grade 3 as per the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE) v5.0) and frequency as compared to placebo at week 12 | Week 12
  Adverse Events severity (as defined by AEs equal or greater than grade 3 as per the National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE) v5.0) and frequency as compared to placebo

SECONDARY OUTCOMES:
Change in the proportion of patients achieving SLE Responder Index-4 (SRI 4) response at week 24 compared to baseline. Another efficacy analysis will be done by comparing subjects treated with Gusacitinib vs. placebo at week 12. | Week 12
  Change in the proportion of patients achieving SLE Responder Index-4 (SRI 4) response at week 24 compared to baseline. Another efficacy analysis will be done by comparing subjects treated with Gusacitinib vs. placebo at week 12. SRI-4 response is defined as:- Reduction of >=4 points from baseline in SLEDAI-2K score- No new BILAG A or no more than 1 new BILAG B disease activity scores- No worsening (defined as an increase of >=0.3 points [10 mm] from baseline) in the Physician s Global Assessment of Disease Activity- Change in SLEDAI-2K total score at week 24

CONTACTS AND LOCATIONS:
Overall Officials: Sarfaraz A Hasni, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001700-AR.html